CLINICAL TRIAL: NCT02460718
Title: ENCOURAGE: Evaluating Community Peer Advisors and Diabetes Outcomes in Rural Alabama
Acronym: ENCOURAGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Monika M. Safford, Professor, Weill Medical College of Cornell University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: T0808270039
Record Dates: First submitted 2015-05-29; First posted 2015-06-02 (Estimated); Last update posted 2016-03-10 (Estimated); Status verified 2016-03

CONDITIONS: Diabetes Mellitus
Keywords: diabetes mellitus; peer support; pragmatic clinical trial
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- control group (No Intervention): Participants received 1-hour group diabetes education class covering diabetes basics, healthy eating, stress reduction, physical activity, social support, and how to get the most out of their doctors visit. Participants also received a diabetes report card showing their Hba1c, blood pressure, ldl cholesterol, and body weight.
- Encourage study (Experimental): Participants in the intervention arm were paired with a peer coach, interacting by telephone weekly for the first 8 weeks and then monthly for a total of 10 months.
  Participants also received 1-hour group diabetes education class covering diabetes basics, healthy eating, stress reduction, physical activity, social support, and how to get the most out of their doctors visit. Participants also received a diabetes report card showing their Hba1c, blood pressure, ldl cholesterol, and body weight.
  Interventions: Behavioral: ENCOURAGE Study

INTERVENTIONS:
Behavioral: ENCOURAGE Study — This intervention tested the effects of a peer coaching program plus brief diabetes education versus brief diabetes education alone on diabetes outcomes.
  Arms: Encourage study

SUMMARY:
It is unclear whether peer coaching is effective in minority populations living with diabetes in hard-to-reach, under resourced areas such as the rural South. We examined the effect of an innovative peer coaching intervention plus brief education vs. brief education alone on diabetes outcomes.

DETAILED DESCRIPTION:
The purpose of this project was to provide robust evidence on the effectiveness of a peer support intervention in improving diabetes outcomes by conducting a group-randomized, controlled implementation trial of a volunteer peer support intervention.

The study had three specific aims:

Aim 1. In Phase I (months 0-8), to perform a qualitative needs assessment with peer advisors and health care providers to inform peer advisor roles and responsibilities (i.e., the intervention) and peer advisor recruitment strategies, curriculum and training; and patient recruitment plans.

Aim 2. Also in Phase I, to pilot our collaboratively developed intervention and, based on pilot test results, to recruit and train peer advisors for the intervention, and begin patient recruitment.

Aim 3. In Phase II (months 9-32), conduct the group randomized implementation trial and evaluate it using the Reach, Effectiveness, Adoption, Implementation, Maintenance (RE-AIM) framework.

ELIGIBILITY:
Inclusion Criteria:

* 19 or older in age, diagnosed with diabetes, under the care of a doctor

Exclusion Criteria:

* not community dwelling, less than 19 years old, pregnant, end-stage medical conditions with limited life expectancy, no access to telephone, does not speak english

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 424 (Actual)
Dates: Start 2009-02; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Glycated hemoglobin (A1c) | Change in A1c in 12 months
  fingerstick, point-of-care a1c test
Blood pressure | Change in blood pressure measure in 12 months
  Measured using digital automated blood pressure monitor
LDL cholesterol | Change in LDL cholesterol in 12 month
  measured using finger stick, spectrophotometer to measure LDL cholesterol
diabetes self-care behaviors questionnaire | Change in diabetes self-care behaviors at 12 months
  aspects of diabetes self-management such as taking medications as directed, self-report of exercise, and eating behaviors
depressive symptoms | change in depressive symptoms at 12 months
  self-report using Patient Health Questionnaire 8 (PHQ8)
quality of life | Change in quality of life measures at 12 months
  self-report using Short form-1 (SF1), and Euroquol (EQ-5D)
patient activation | change in patient activation in 12 months
  self-report using the 13 item Patient Activation Measure (PAM13)

SECONDARY OUTCOMES:
body mass index | change in BMI in 12 months
  weight measured using digital scale, height measured using stadiometer
diabetes knowledge | change in diabetes knowledge in 12 months
  assessed using the Spoken Knowledge in Low Literacy in Diabetes Scale
trust in physicians | change in trust in physicians in 12 months
  assessed using the Trust in Physicians Scale
composite measure of healthcare utilization | Change in health care utilization in 12 months
  self-report by participant, number of times utilized healthcare services

IPD SHARING:
Plan to Share IPD: No
Data will stay at UAB

REFERENCES:
- [Derived] Cherrington AL, Khodneva Y, Richman JS, Andreae SJ, Gamboa C, Safford MM. Impact of Peer Support on Acute Care Visits and Hospitalizations for Individuals With Diabetes and Depressive Symptoms: A Cluster-Randomized Controlled Trial. Diabetes Care. 2018 Dec;41(12):2463-2470. doi: 10.2337/dc18-0550. Epub 2018 Oct 29. PMID 30373734